CLINICAL TRIAL: NCT01131494
Title: Dysphagia Therapy for Parkinson's Disease: the Role of the Oral Motor Exercises
Brief Title: Swallowing Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Natalie Argolo Pereira Ponte, PhD Student, Federal University of Bahia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 249/2008
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-10

CONDITIONS: Parkinson's Disease; Deglutition Disorders; Voice Disorders
Keywords: Parkinson's disease; Dysphagia; Treatment
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders; Voice Disorders | interventions — Deglutition; Respiration; Phonation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Swallowing exercises (Experimental)
  Interventions: Other: Motor exercises for swallowing, breathing and phonation

INTERVENTIONS:
Other: Motor exercises for swallowing, breathing and phonation — This exercises aimed to increase strength and range of motion of mouth, larynx and pharynx structures. All patients made sustained vowel phonation of /a/, pushing plosive phonemes /pa/, /ta/, /ka/ in a forceful manner, suction of wet gauze, swallowing with tongue hold and modified supraglottic maneuver, in ten repetitions, ascending and descending gliding phonation of vowel /a/ and /u/, five repetitions of each vowel, and tongue rotation in oral vestibule, 3 series of 5 repetitions to each side. Patients underwent oral motor exercises twice a day, five days a week, for five weeks.

SUMMARY:
Dysphagia in Parkinson's disease(PD) is common and its presence is related to motor and sensory abnormalities, and incoordination between swallowing and breathing. Despite harming as respiratory infections and increased risk of death, treatment of this condition remains uncertain. This study aims to evaluate the effect of oral motor exercises on the swallowing dynamics and quality of life of dysphagic Parkinson's disease patients. This study is an open trial, self-paired and blinded to the examiner. The participants will perform oropharyngeal exercises for five weeks and will be evaluated before and after intervention by swallowing videofluoroscopy and questionnaires about quality of life in dysphagia (SWAL-QOL).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson disease
* Complaint of dysphagia

Exclusion Criteria:

* Hoehn and Yahr stage 5
* Other neurological conditions
* Therapy for swallowing in the last 3 months
* Cognitive disorders
* Psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Caline Nóbrega, PhD, Study Chair — Federal University of Bahia
Locations (1):
- Federal University of Bahia, Salvador, Estado de Bahia, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients from Movement Disorders Ambulatory of Federal University of Bahia in Brazil with idiopathic Parkinson disease (IPD) and complaint of dysphagia, from March 2009 to June 2010, were invited to participate.
Pre-assignment Details: Patients with severe dysphagia who needed others interventions (for example: management of food consistency, alternative way of feeding) were excluded. During the study, subjects with absence in three sessions of exercises were excluded from the study and sent to Ambulatory of Speech and Deglutition Disorders at Federal University of Bahia.
Groups:
- Swallowing Exercise Group: One group made swallowing exercises for five weeks. This group was compared before and after the study.
Period: Overall Study
Arm/Group | Swallowing Exercise Group
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Swallowing Exercise Group
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 60.12 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Region of Enrollment [Number; unit: participants]
  Brazil | 17

OUTCOME MEASURES:

1. Secondary Outcome: Quality of Life
Description: Measured by the Swal-qol (Quality of life in Swallowing disorders). In this questionnaire the score range from 0 to 100 and higher scores is better quality of life.
Time Frame: five weeks
Measure: Median (Inter-Quartile Range); unit: scores in a scale
Groups:
- Pre-intervention Measure: Measurements of the group made before begin intervention.
- Post-intervention Measure: Measurements of the group made after the intervention.
Arm/Group | Pre-intervention Measure | Post-intervention Measure
Number analyzed (Participants) | 15 | 15
scores in a scale | 64.33 [40.05 to 79.8] | 70.58 [47.72 to 77.13]

2. Primary Outcome: Oropharyngeal Swallowing Score
Description: Based on videofluoroscopy, were awarded points for the swallowing events according to their clinical relevance. The sum of these points results in the OSP (Oropharyngeal Swallowing Score), so that higher scores signify greater impairment in swallowing. OSP-score range from 0 to 243.5. This tool is being validated for that group.
Time Frame: five weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pre-intervention Measure | Post-intervention Measure
Number analyzed (Participants) | 15 | 15
Scores on a scale | 22.15 (9.36) | 21.93 (12.81)

ADVERSE EVENTS:
Time Frame: Adverse event was not collected after end of study.
Description: No formal tool to collect adverse event was used because there is no report that oral exercise can cause adverse event.
Arm/Group | Swallowing Exercise Group
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
There was a delay because of faulty equipment that performs videofluoroscopy of swallowing.

Study limitations include small number of participants and no comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No